CLINICAL TRIAL: NCT06876402
Title: Assessment of the Prevalence and Prognostic Value of Gene Molecular Alterations and Association With Clinicopathological Factors in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Gene Molecular Alterations as Disease Prognostic Markers in Patients With Non-small Cell Lung Cancer (NSCLC)
Acronym: GEMA-proN
Status: Active, not recruiting | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE_2TR/13
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: NSCLC; Non-small cell lung cancer; Early stage non-small cell lung cancer; Metastatic non-small cell lung cancer; Mutations; Copy number alterations; Translocations; CNA; PD-L1 expression; Tumor infiltrating lymphocytes; TILs; Pathogenic single nucleotide variants
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extraction from formalin fixed paraffin-embeded tissue (FFPE). 2 blocks, 5 sections per patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with histologically confirmed diagnosis of non-small cell lung cancer (NSCLC).: Assessment of tumor molecular profile in patients with histologically confirmed early stage or metastatic non-small cell lung cancer (NSCLC).
  Identification of gene somatic alterations including single nucleotide variants (SNVs), small insertions and deletions (indels), copy number alterations (CNAs), and rearrangements with the use of next generation sequencing (NGS) with a custom tumor profile gene assay developed by NIPD Genetics.

SUMMARY:
GEMA-proN is an observational, multicenter, single cohort, retrospective clinical trial. The aim of the trial is to assess the prevalence, and prognostic value of genetic molecular alterations and investigate correlations with clinicopathological features in unselected patients with histologically confirmed non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This a non- interventional, multicenter, retrospective one arm trial assessing patients with histologically confirmed diagnosis of non-small cell lung cancer (NSCLC). Patients received treatment in 18 Hellenic Cooperative Oncology Group (HeCOG)- affiliated centers in Greece between 2000 and 2020. Molecular genetic alterations, including single nucleotide variants, copy number alterations, and translocations, are detected with next generation sequencing using the ForeSENTIA® NSCLC panel developed by NIPD Genetics. The aim of the trial is to assess the prevalence and prognostic value of molecular alterations in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above.
* Histologically confirmed non-small cell lung cancer (NSCLC).
* Adequate, and suitable tissue for the testing of somatic genetic alterations.

Exclusion Criteria:

- Patients with personal medical history of malignancy, other than non-small cell lung cancer (NSCLC), with the exclusion of completely resected non-melanoma skin cancers, in situ carcinomas of the cervix uteri, in situ bladder carcinomas, in situ ductal breast carcinoma, and other cancers treated with curative intent with no evidence of disease recurrence for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-small cell lung cancer (NSCLC) regardless of disease stage, between 2000 and 2020, who received treatment in 18 Hellenic Cooperative Oncology Group (HeCOG)- affiliated centers in Greece.
  Variables under investigation;
  * ECOG performance status (categorical),
  * Sex (categorical)
  * Age (continuous)
  * Smoking status (categorical)
  * Histology type (categorical)
  * Stage (categorical)
  * Type of surgery in resected disease (categorical)
  * Pathogenic/ likely pathogenic SNVs (categorical)
  * CNAs (categorical)
  * Translocations (categorical)
  * Co-mutations (categorical)
  * PD-L1 expression (categorical)
  * TILs expression (categorical)
  * Immunotherapy in the 1st line setting (categorical)
  * Overall survival (OS) (continuous)
  * PFS (progression-free survival)
  * DFS (disease-free survival)
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
OS (overall survival) in whole cohort. | Through study completion, 3 years.
  Overall survival is defined from the date of initial diagnosis until death or last contact.

SECONDARY OUTCOMES:
Progression-free survival (PFS) in patients who received 1st line treatment for metastatic non-small cell ling cancer (NSCLC). | Through study completion, 3 years.
  Progression-free survival is defined from the date of 1st line treatment initiation until the date of radiologically confirmed disease progression (PD), following 1st line treatment.
Recurrence-free survival (RFS) in patients who underwent surgical treatment for non-small cell lung cancer (NSCLC). | Through study completion, 3 years.
  Recurrence-free survival is defined from the date of initial surgical diagnosis until the date of radiologically confirmed disease recurrence, following surgical resection.

OTHER OUTCOMES:
Prevalence of somatic gene alterations. | Through study completion, 3 years.
  Assessment of the prevalence of detected pathogenic/ likely pathogenic single nucleotide variants (SNVs), copy number alterations (CNAs), translocations, and co-mutations.
Prognostic value of assessed somatic gene molecular alterations. | Through study completion, 3 years
  Assessment of the prognostic value of detected pathogenic/ likely pathogenic single nucleotide variants (SNVs), copy number alterations (CNAs), translocations, and co-mutations.
Prognostic value of assessed PD-L1 expression. | Through study completion, 3 years.
  Assessment of the prognostic value of PD-L1 expression.
Prognostic value of tumor-infiltrating lymphocytes (TILs). | Through study completion, 3 years.
  Assessment of the prognostic value of tumor-infiltrating lymphocytes (TILs).

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Cooperative Oncology Group (HeCOG), Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular profiling of lung adenocarcinoma. Nature. 2014 Jul 31;511(7511):543-50. doi: 10.1038/nature13385. Epub 2014 Jul 9. PMID 25079552
- [Background] Cancer Genome Atlas Research Network. Comprehensive genomic characterization of squamous cell lung cancers. Nature. 2012 Sep 27;489(7417):519-25. doi: 10.1038/nature11404. Epub 2012 Sep 9. PMID 22960745
- [Background] Skoulidis F, Heymach JV. Co-occurring genomic alterations in non-small-cell lung cancer biology and therapy. Nat Rev Cancer. 2019 Sep;19(9):495-509. doi: 10.1038/s41568-019-0179-8. Epub 2019 Aug 12. PMID 31406302
- [Background] Hendry S, Salgado R, Gevaert T, Russell PA, John T, Thapa B, Christie M, van de Vijver K, Estrada MV, Gonzalez-Ericsson PI, Sanders M, Solomon B, Solinas C, Van den Eynden GGGM, Allory Y, Preusser M, Hainfellner J, Pruneri G, Vingiani A, Demaria S, Symmans F, Nuciforo P, Comerma L, Thompson EA, Lakhani S, Kim SR, Schnitt S, Colpaert C, Sotiriou C, Scherer SJ, Ignatiadis M, Badve S, Pierce RH, Viale G, Sirtaine N, Penault-Llorca F, Sugie T, Fineberg S, Paik S, Srinivasan A, Richardson A, Wang Y, Chmielik E, Brock J, Johnson DB, Balko J, Wienert S, Bossuyt V, Michiels S, Ternes N, Burchardi N, Luen SJ, Savas P, Klauschen F, Watson PH, Nelson BH, Criscitiello C, O'Toole S, Larsimont D, de Wind R, Curigliano G, Andre F, Lacroix-Triki M, van de Vijver M, Rojo F, Floris G, Bedri S, Sparano J, Rimm D, Nielsen T, Kos Z, Hewitt S, Singh B, Farshid G, Loibl S, Allison KH, Tung N, Adams S, Willard-Gallo K, Horlings HM, Gandhi L, Moreira A, Hirsch F, Dieci MV, Urbanowicz M, Brcic I, Korski K, Gaire F, Koeppen H, Lo A, Giltnane J, Rebelatto MC, Steele KE, Zha J, Emancipator K, Juco JW, Denkert C, Reis-Filho J, Loi S, Fox SB. Assessing Tumor-Infiltrating Lymphocytes in Solid Tumors: A Practical Review for Pathologists and Proposal for a Standardized Method from the International Immuno-Oncology Biomarkers Working Group: Part 2: TILs in Melanoma, Gastrointestinal Tract Carcinomas, Non-Small Cell Lung Carcinoma and Mesothelioma, Endometrial and Ovarian Carcinomas, Squamous Cell Carcinoma of the Head and Neck, Genitourinary Carcinomas, and Primary Brain Tumors. Adv Anat Pathol. 2017 Nov;24(6):311-335. doi: 10.1097/PAP.0000000000000161. PMID 28777143
- [Background] Tuminello S, Sikavi D, Veluswamy R, Gamarra C, Lieberman-Cribbin W, Flores R, Taioli E. PD-L1 as a prognostic biomarker in surgically resectable non-small cell lung cancer: a meta-analysis. Transl Lung Cancer Res. 2020 Aug;9(4):1343-1360. doi: 10.21037/tlcr-19-638. PMID 32953509